CLINICAL TRIAL: NCT05574829
Title: Assessment of Neural Pressure Support Assisted Ventilation and Non-invasive Estimation of Transpulmonary Pressure in Spontaneous Ventilation Modes
Brief Title: Neural Pressure Support and Non-invasive Estimation of Transpulmonary Pressure in Spontaneous Ventilation Modes
Acronym: EADITRAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Maquet Critical Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: EADITRAP
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients under pressure support ventilation: Patients under assisted mechanical ventilation monitored with esophageal manometry and electrical activity of the diaphragm
  Interventions: Device: Esophageal manometry and monitoring of electrical activity of the diaphragm

INTERVENTIONS:
Device: Esophageal manometry and monitoring of electrical activity of the diaphragm — Esophageal manometry and monitoring of electrical activity of the diaphragm

SUMMARY:
The transition from controlled mechanical ventilation to assisted ventilation is one of the most complex and compromised phases of the ventilatory management during mechanical ventilation, affected by factors such as:

* Asynchronies, due to patient-respirator dis-synchrony in ins- and expiratory neural and mechanical times, as well as inadequate levels of assistance.
* Risks of self-induced lung injury resulting from uncontrolled increases in transpulmonary pressure when high inspiratory efforts are combined with inappropriate levels of inspiratory pressure assistance.

Current monitoring of assisted ventilation is complex and not well resolved by most conventional ventilators. Asynchronies are difficult to monitor with the pressure or flow/time curves present in conventional ventilators requiring an advanced level of expertise. Measurements of the patient's muscular effort and therefore of transpulmonary pressure, requires the use of esophageal manometry with cumbersome handling and interpretation.

NAVA (Neurally Adjusted Ventilatory Assist) is a ventilator mode that uses electrical activity of the diaphragm (EAdi), monitored via a modified nasogastric feeding catheter, to control and assist the respiratory cycle by the ventilator. Recently, a "hybrid" mode between the conventional pressure support assisted mode (PSV) and NAVA called Neural-Pressure Support Ventilation (N-PSV) has been developed. This mode uses a neural trigger based on the EAdi to match the patient's and ventilator's in- and expiratory time, but unlike NAVA, assisting in the same way as in pressure support. In addition the EAdi allows to assess the extent to which the patient's muscle strength contributes to the patient-ventilator breath (PVBC), and it has recently been suggested that on the basis of PVBC it may also be possible to directly estimate the patient's transpulmonary pressure (PL).

Hypothesis:

1. EAdi allows direct estimation of PL during the assisted ventilation phase without the need of an oesophageal pressure balloon.
2. N-PSV can provide advantages over PSV by better matching ventilator and patient respiratory cycle times, thus reducing the risk of asynchronies.

DETAILED DESCRIPTION:
Consenting participants will be simultaneously monitored with a 8French EAdi catheter (to measure the electrical activity of the diaphragm) and a 15French nasogastric catheter with an oesophageal balloon to measure oesophageal manometry during the 120 min of the total study period.

After confirming correct positioning and measurement of both catheters participants will be submitted to the following protocol:

Baseline ventilation in pressure support ventilation during 30 min Baseline ventilation in neural-pressure support ventilation during 30 min Under-assistance in neural pressure support ventilation reducing the baseline level of pressure support by 50% (with a minimum of 5 cmH2O) during 30 min Over-assistance in neural pressure support ventilation by increasing the baseline level of pressure by 50% during 30 min.

The sequence of the last two steps will be randomly determined. After completing the protocol the EAdi catheter will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mechanically assisted ventilation
* Patients with a nasogastric catheter
* Obtained informed consent
* Clinical stability, defined as:

  * Low ventilatory support requirement: FiO2 (Fraction of inspired oxygen) ≤ 0.5; PEEP (positive end-expiratory pressure) ≤ 10 cmH2O (up to 12 cmH2O for patients with a body mass index ≥ 30 kg/m2).
  * Haemodynamic stability: a)low vasopressor requirement: Noradrenaline ≤ 0.2 microg/kg/min; b)Mean blood pressure ≥ 60 mmHg; c)No new arrhythmias.

Exclusion Criteria:

* Presence of Contraindications for the insertion of a nasogastric tube: oesophageal pathology. Coagulopathy, bleeding diathesis
* Clinical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients under assisted mechanical ventilation with spontaneous breathing and adequate respiratory drive.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of asynchronies | 60 minutes
  Asynchrony index
Estimation of transpulmonary pressure | 90 minutes
  Evaluation of a new method for measuring transpulmonary pressure based on the electrical activity of the diaphragm

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No